CLINICAL TRIAL: NCT00824148
Title: Use of Real-time Continuous Glucose Monitoring System to Control Blood Glucose in Patients With Type 1 Diabetes Mellitus
Brief Title: Use of Real-time Continuous Glucose Monitoring System in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4.2008.1607; 19637 (Other: NSD)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Real-time glucose monitoring system; HbA1c; Quality of life; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time glucose monitoring (Experimental): Use of Guardian REAL-Time Continuous Glucose Monitoring System, (Medtronic Minimed, Northridge, CA) for 1 month, followed by observation for 2 months.
  Interventions: Device: Guardian REAL-Time Continuous Glucose Monitoring System
- Self-monitoring of plasma glucose (Active Comparator): Conventional self-monitoring of plasma glucose by finger-prick sampling for 1 month, followed by 1 month observation.
  Interventions: Other: Conventional self-monitoring of plasma glucose

INTERVENTIONS:
Device: Guardian REAL-Time Continuous Glucose Monitoring System — One group will use the glucose monitoring system for 1 month
  Arms: Real-time glucose monitoring
Other: Conventional self-monitoring of plasma glucose — Finger prick blood glucose measurements
  Arms: Self-monitoring of plasma glucose

SUMMARY:
The purpose of this study is to determine whether a real-time continuous glucose monitoring system is able to improve HbA1c in patients suffering from type 1 diabetes compared to conventional finger prick glucose measurements. In addition it will investigate whether number of episodes with serious hypoglycemia is changed in those same patients, and whether quality of life (health status and treatment satisfaction) increases.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes Mellitus, Type 1 > 3 years.
2. For practical reasons patients should live in Trondheim, Malvik, Melhus or Klæbu.
3. Level of HbA1c (measured by DCA 2000) between 7 and 10 % and/or experience blood glucose < 3 mmol/L (verified by finger-prick measurement) at least once a week and/or at least one episode with serious hypoglycemia the previous half a year.(Defined as need of help from others)
4. Only patients who use insulin pumps or multi-injection regime (=3 daily injections with short term acting insulin or insulin analogue + at lest one daily injection with NPH-insulin or long term acting insulin analogue.

Exclusion Criteria:

1. Patients with other diseases such as untreated hypothyroidism, adrenal gland failure, celiac disease, renal failure, unstable coronary heart disease, serious psychiatric disorder, or mental retardation.
2. Patients who are not able to learn how to use the continuous glucose monitoring system given a reasonable amount of effort.
3. Patients who are not able to do the glucose measurements, insulin dose change and diary notes which the study demands.
4. Unsuited for participating from any other cause.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Level of HbA1c concentration | 1 and 3 months post intervention.

SECONDARY OUTCOMES:
Quality of life assessed by SF-36, DTSQs and DTSQc | 1 and 3 months post intervention
Number of hypoglycemic events | 1 and 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kristian J Fougner, MD, Principal Investigator — Departement of Endocrinology St. Olavs Hospital
Locations (1):
- Department of Endocrinology, St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Langeland LB, Salvesen O, Selle H, Carlsen SM, Fougner KJ. Short-term continuous glucose monitoring: effects on glucose and treatment satisfaction in patients with type 1 diabetes mellitus; a randomized controlled trial. Int J Clin Pract. 2012 Aug;66(8):741-747. doi: 10.1111/j.1742-1241.2012.02947.x. PMID 22805265